CLINICAL TRIAL: NCT06486337
Title: A Single-arm, Multi-center, Prospective Clinical Study of Mitoxantrone Hydrochloride Liposome Injection-based CMOP±R Regimen in the Treatment of Newly Diagnosed Non-Hodgkin's Lymphoma
Brief Title: CMOP±R in the Treatment of Untreated Non-Hodgkin's Lymphoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-DED-NHL-K03
Record Dates: First submitted 2024-06-16; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-05

CONDITIONS: NHL
Keywords: newly diagnosed non-Hodgkin's lymphoma; Mitoxantrone hydrochloride liposome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CMOP±R (Experimental): All enrolled patients. All patient who signed the consent form for participation to the study.
  Interventions: Drug: CMOP±R

INTERVENTIONS:
Drug: CMOP±R — Drug: Mitoxantrone hydrochloride liposome Mitoxantrone hydrochloride liposome (18 mg/m^2) on day 1, every 4 weeks; Drug: Cyclophosphamide Cyclophosphamide(750 mg/m^2) on day 1, every 4 weeks; Drug: Vincristine Vincristine (1.4mg/ m2，Max dose 2mg) will be administered on day 1(Or at the discretion of the investigator, use other vinblastine drugs with the same mechanism, such as vindesine 2-3 mg/m2 on day 1), every 4 weeks; Drug: Prednisone Prednisone (100 mg) will be taken orally from day 1-5(Or equivalent dose of dexamethasone at 15mg), every 4 weeks; Drug: Rituximab Rituximab (375mg/m^2) on day 0, every 4 weeks, only with CD20-positive lymphomas are evaluated by the investigator.

SUMMARY:
This is a prospective, single arm, multicenter study to evaluate the safety and efficacy of CMOP±R in patients with newly diagnosed non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
This is a single-arm, open label, multi-center clinical study to evaluate the safety and efficacy of mitoxantrone hydrochloride liposome in combination with Cyclophosphamide, Vincristine, Prednisone and/or Rituximab(CMOP±R) in patients with newly diagnosed non-Hodgkin's lymphoma. Mitoxantrone hydrochloride liposome will be given on day 1 at dose of 18 mg/m2 and be combined with cyclophosphamide, vincristine, prednisone and/or Rituximab. Each cycle consists of 28 days. A maximum of 8 cycles(6×CMOP±R+2×R) of therapy are planned.

ELIGIBILITY:
Inclusion Criteria:

* Patients fully understand this study, voluntarily participate and sign the informed consent (ICF);
* Age: 18-75 years old;
* Expected survival time ≥ 3 months;
* Histopathologically diagnosed newly diagnosed non-Hodgkin's lymphoma;
* Must have at least one evaluable or measurable lesion that meets the Lugano 2014 criteria: lymph node lesions, measurable lymph nodes must have a long diameter >1.5cm; non-lymph node lesions, measurable extranodal lesions must have a long diameter >1.0cm;
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0-2.
* Bone marrow function: Absolute neutrophil count (ANC) ≥1.5×10^9/L, Platelet count (PLT) ≥75×10^9/L, Hemoglobin(HB)≥ 80 g/L(Restriction may be relaxed in patients with bone marrow involvement, Absolute neutrophil count (ANC) ≥1.0×10^9/L, Platelet count (PLT) ≥50×10^9/L, Hemoglobin(HB)≥ 75g/L);
* Liver and kidney function: serum creatinine ≤ 1.5 times the upper limit of normal value; AST and ALT ≤ 2.5 times the upper limit of normal value (for patients with liver invasion ≤ 5 times the upper limit of normal value); total bilirubin ≤ 1.5 times the upper limit of normal value (for patients with liver invasion ≤ 3 times the upper limit of normal value);

Exclusion Criteria:

* Subjects have previously received anthracyclic drug pretreatment;
* Hypersensitivity to any study drug or its components;
* Uncontrollable systemic diseases (such as advanced infection, uncontrollable hypertension, diabetes, etc.);
* Heart function and disease meet one of the following conditions: a) long QTc syndrome or QTc interval >480 ms; b) complete left bundle branch block, grade II or III atrioventricular block; c) Serious and uncontrolled arrhythmias requiring drug treatment; d) New York Heart Association grade ≥ III; e) Cardiac ejection fraction (LVEF) lower than 50%;f) A history of myocardial infarction, unstable angina pectoris, severe unstable ventricular arrhythmia or any other arrhythmia requiring treatment, a history of clinically serious pericardial disease, or ECG evidence of acute ischemia or active conduction system abnormalities within 6 months before recruitment.
* Active hepatitis B and C infection (positive hepatitis B virus surface antigen and more than 1x10^3 copies/mL of hepatitis B virus DNA; more than 1x10^3 copies/mL of hepatitis C virus RNA);
* Human immunodeficiency virus (HIV) infection (positive HIV antibody);
* Suffering from other malignant tumors in the past or at the same time (except for effectively controlled non-melanoma skin basal cell carcinoma, breast/cervix carcinoma in situ, and other malignant tumors that have been effectively controlled without treatment in the past five years);
* Suffering from primary or secondary central nervous system (CNS) lymphoma or a history of CNS lymphoma at the time of recruitment;
* Pregnant and lactating women and patients of childbearing age who are unwilling to take contraceptive measures;
* Other researchers judge not to Eligibility to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Estimated)
Dates: Start 2024-07-10 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Complete Response Rate (CRR) | 3 years
  Response is assessed according to the 2014 lugano criteria.Percentage of participants with complete response was determined on 2014 Lugano criteria.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | 3 years
  Response is assessed according to the 2014 lugano criteria.The total percentage of patients with complete response（CR ）and partial response（PR).
Progression-Free-Survival (PFS) | 3 years
  From the time subjects were enrolled to the time of disease progression (in any way) or death from any cause.Progression-free survival (PFS) was analyzed using Kaplan-Meier method, and 95% bilateral confidence intervals were calculated.
Duration of Response (DOR) | 3 years
  The time between meeting the criteria for treatment effectiveness (first recorded complete or partial response) and the first clear recurrence or progression.Duration of response (DoR) was analyzed using Kaplan-Meier method, and 95% bilateral confidence intervals were calculated.
Overall survival (OS) | 3 years
  From the date of inclusion to date of death, irrespective of cause.Overall survival (OS) was analyzed using Kaplan-Meier method, and 95% bilateral confidence intervals were calculated.
Progression of disease within 2 years(POD24) | 3 years
  The rate of patients with disease progression within 24 months of receiving first-line treatment at the start of enrollment.
Treatment-emergent adverse events (TEAEs) | From the initiation of the first dose to 28 days after the last dose
  The safety of the drug was evaluated by NCI-CTC AE 5.0 standard.Hematologic and non-hematologic toxicity.To identify the incidence of TEAEs with NCI-CTC AE 5.0 standard.
Changes in cardiac safety indicators | 3 years
  The change value of LVEF% from baseline, and its mean, median, standard deviation, maximum and minimum values were statistically described.

CONTACTS AND LOCATIONS:
Overall Officials: Haiwen Huang, Principal Investigator — The First Affiliated Hospital of Soochow University, Suzhou, China

IPD SHARING:
Plan to Share IPD: No